CLINICAL TRIAL: NCT00080301
Title: A Phase III Trial of Novel Epothilone BMS-247550 Plus Capecitabine Versus Capecitabine Alone in Patients With Advanced Breast Cancer Previously Treated With or Resistant to an Anthracycline and Who Are Taxane Resistant
Brief Title: Novel Epothilone Plus Capecitabine Versus Capecitabine Alone in Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA163-046
Record Dates: First submitted 2004-03-26; First posted 2004-03-30 (Estimated); Results first posted 2009-08-17 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer; Metastases
Keywords: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — ixabepilone; Capecitabine; Epothilones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Ixabepilone + Capecitabine
- B (Active Comparator)
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Ixabepilone + Capecitabine — Ixabepilone - Intravenous Solution, IV 40mg/m², Day 1 every 21 days, Until progression/unacceptable toxicity
  Capecitabine (Active Comparator) - Tablet, Oral, 2000 mg/m², Bid Days 1-14 every 21 days, Until progression/unacceptable toxicity
  Other Names: BMS-247550; IXEMPRA; Epothilone
  Arms: A
Drug: Capecitabine — Tablet, Oral, 2500 mg/m², Bid Days 1-14 every 21 days, Until progression/unacceptable toxicity
  Arms: B

SUMMARY:
The purpose of this clinical research study is to learn if BMS-247550 added to the approved therapy of capecitabine is better than capecitabine alone in shrinking or slowing the growth of the cancer in women with metastatic breast cancer who are resistant to taxane and received anthracycline chemotherapy. The safety of this treatment will also be studied.

ELIGIBILITY:
* Patients must have received either 2 or 3 prior chemotherapy regimens including adjuvant or neoadjuvant therapy.
* Prior treatment must have included both an anthracycline (i.e., doxorubicin or epirubicin) and a taxane (i.e., paclitaxel or docetaxel).
* Patients must have received a minimum cumulative dose of anthracycline or must be resistant to an anthracycline.
* Patients must be resistant to taxane therapy.
* Patients may not have any history of brain and/or leptomeningeal metastases.
* Patients may not have CTC Grade 2 or greater neuropathy (motor or sensory).
* Patients may have not have had prior treatment with an epothilone and/or capecitabine (i.e., Xeloda)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Actual)
Dates: Start 2003-09; Primary Completion 2006-11 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (127):
- United States (32):
  - Local Institution, Little Rock, Arkansas
  - Local Institution, San Francisco, California
  - Local Institution, Vallejo, California
  - Local Institution, Denver, Colorado
  - Local Institution, Hartford, Connecticut
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Orlando, Florida
  - Local Institution, Baltimore, Maryland
  - Local Institution, Burlington, Massachusetts
  - Local Institution, Jackson, Mississippi
  - Local Institution, Columbia, Missouri
  - Local Institution, Kansas City, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution, Omaha, Nebraska
  - Local Institution, Livingston, New Jersey
  - Local Institution, New Brunswick, New Jersey
  - Local Institution, Albuquerque, New Mexico
  - Local Institution, New York, New York
  - Local Institution, Columbus, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Tulsa, Oklahoma
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Columbia, South Carolina
  - Local Institution, Greenville, South Carolina
  - Local Institution, Knoxville, Tennessee
  - Local Institution, Nashville, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Ogden, Utah
  - Local Institution, Burlington, Vermont
  - Local Institution, Tacoma, Washington
  - Local Institution, Morgantown, West Virginia
- Argentina (11):
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Haedo, Buenos Aires
  - Local Institution, La Plata, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, Pilar, Buenos Aires
  - Local Institution, Quilmes, Buenos Aires
  - Local Institution, Lanús, BuenosAires
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, Córdoba
  - Local Institution, Neuquén
  - Local Institution, Santa Fe
- Belgium (4):
  - Local Institution, Edegem
  - Local Institution, Ghent
  - Local Institution, Leuven
  - Local Institution, Liège
- Brazil (8):
  - Local Institution, Fortaleza, Ceará
  - Local Institution, Belo Horizonte, Mina Gerais
  - Local Institution, Curitiba, Paraná
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Jaú, São Paulo
  - Local Institution, Santo André, São Paulo
  - Local Institution, Sao Paulo - Sp, São Paulo
  - Local Institution, São Paulo
- Canada (4):
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Oshawa, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
- China (8):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Jinan, Shandong
  - Local Institution, Beijing, Shanghai Municipality
  - Local Institution, Xi’an, Shanxi
  - Local Institution, Beijing
  - Local Institution, Shanghai
- France (15):
  - Local Institution, Angers
  - Local Institution, Avignon
  - Local Institution, Bayonne
  - Local Institution, Besançon
  - Local Institution, Bobigny
  - Local Institution, Bordeaux
  - Local Institution, Clermont-Ferrand
  - Local Institution, Lyon
  - Local Institution, Nantes
  - Local Institution, Nice
  - Local Institution, Saint-Brieuc
  - Local Institution, Saint-Cloud
  - Local Institution, Saint-Herblain
  - Local Institution, Strasbourg
  - Local Institution, Toulouse
- Germany (3):
  - Local Institution, Berlin
  - Local Institution, Duisburg
  - Local Institution, Erlangen
- Greece (2):
  - Local Institution, Athens
  - Local Institution, Thessaloniki
- Hungary (4):
  - Local Institution, Budapest
  - Local Institution, Debrecen
  - Local Institution, Győr
  - Local Institution, Pécs
- Italy (4):
  - Local Institution, Brescia
  - Local Institution, Candiolo (To)
  - Local Institution, Forlì
  - Local Institution, San Giovanni Rotondo
- Malaysia (2):
  - Local Institution, Kampung Baharu Nilai, Negeri Sembilan
  - Local Institution, Kuala Lumpur
- Mexico (5):
  - Local Institution, Acapulco de Juárez, Guerrero
  - Local Institution, Mérida, Yucatán
  - Local Institution, Chihuahua City
  - Local Institution, Distrito Federal
  - Local Institution, San Luis Potosí City
- Local Institution, Lima, Peru
- Philippines (3):
  - Local Institution, Manila
  - Local Institution, Quezon
  - Local Institution, Quezon City
- Poland (2):
  - Local Institution, Gdansk
  - Local Institution, Opole
- South Korea (2):
  - Local Institution, Incheon
  - Local Institution, Seoul
- Spain (5):
  - Local Institution, Barcelona
  - Local Institution, Girona
  - Local Institution, Madrid
  - Local Institution, Valencia
  - Local Institution, Zaragoza
- Sweden (2):
  - Local Institution, Gothenburg
  - Local Institution, Stockholm
- Taiwan (2):
  - Local Institution, Tainan
  - Local Institution, Taipei
- Local Institution, Bangkok, Thailand
- United Kingdom (7):
  - Local Institution, Bristol, Avon
  - Local Institution, Chelmsford, Essex
  - Local Institution, London, Greater London
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Sheffield, South Yorkshire
  - Local Institution, Guildford, Surrey
  - Local Institution, Newcastle upon Tyne, Tyne and Wear

REFERENCES:
- [Result] Thomas ES, Gomez HL, Li RK, Chung HC, Fein LE, Chan VF, Jassem J, Pivot XB, Klimovsky JV, de Mendoza FH, Xu B, Campone M, Lerzo GL, Peck RA, Mukhopadhyay P, Vahdat LT, Roche HH. Ixabepilone plus capecitabine for metastatic breast cancer progressing after anthracycline and taxane treatment. J Clin Oncol. 2007 Nov 20;25(33):5210-7. doi: 10.1200/JCO.2007.12.6557. Epub 2007 Oct 29. PMID 17968020
- [Derived] Vahdat LT, Vrdoljak E, Gomez H, Li RK, Bosserman L, Sparano JA, Baselga J, Mukhopadhyay P, Valero V. Efficacy and safety of ixabepilone plus capecitabine in elderly patients with anthracycline- and taxane-pretreated metastatic breast cancer. J Geriatr Oncol. 2013 Oct;4(4):346-52. doi: 10.1016/j.jgo.2013.07.006. Epub 2013 Aug 23. PMID 24472478
- [Derived] Jassem J, Fein L, Karwal M, Campone M, Peck R, Poulart V, Vahdat L. Ixabepilone plus capecitabine in advanced breast cancer patients with early relapse after adjuvant anthracyclines and taxanes: a pooled subset analysis of two phase III studies. Breast. 2012 Feb;21(1):89-94. doi: 10.1016/j.breast.2011.09.003. Epub 2011 Sep 21. PMID 21937232
- [Derived] Roche H, Conte P, Perez EA, Sparano JA, Xu B, Jassem J, Peck R, Kelleher T, Hortobagyi GN. Ixabepilone plus capecitabine in metastatic breast cancer patients with reduced performance status previously treated with anthracyclines and taxanes: a pooled analysis by performance status of efficacy and safety data from 2 phase III studies. Breast Cancer Res Treat. 2011 Feb;125(3):755-65. doi: 10.1007/s10549-010-1251-y. Epub 2010 Dec 3. PMID 21128114

RESULTS

PARTICIPANT FLOW:
Groups:
- Ixabepilone + Capecitabine: Ixabepilone 40 mg/m2 administered as a 3-hour intravenous (IV) infusion on Day 1 of each 21-day cycle, plus oral capecitabine 1000 mg/m2 twice a day (BID) x 14 days
- Capecitabine: Capecitabine 1250 mg/m2 BID x 14 days
Period: Overall Study
Arm/Group | Ixabepilone + Capecitabine | Capecitabine
Started | 375 | 377
Never Treated | 5 | 10
Still on Treatment | 0 | 1
Completed | 370 (Participants who are off treatment) | 366 (Participants who are off treatment)
Not Completed | 5 | 11
Not completed — Randomized but Never Treated | 5 | 10
Not completed — Still on Treatment as of CSR date | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixabepilone + Capecitabine | Capecitabine | Total
Number analyzed (Participants) | 375 | 377 | 752
Age, Customized [Number; unit: participants]
  <65 years | 336 | 322 | 658
  >= 65 years | 39 | 54 | 93
  <50 years | 135 | 145 | 280
  >= 50 years | 240 | 231 | 471
  Unknown | 0 | 1 | 1
Age, Continuous [Median (Full Range); unit: years] | 53.0 [25.0 to 76.0] | 52.0 [25.0 to 79.0] | 53.0 [25.0 to 79.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 375 | 376 | 751
  Male | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 83 | 87 | 170
  Black or African American | 11 | 11 | 22
  White | 257 | 247 | 504
  Other | 23 | 32 | 55
Disease Sites [Number; unit: participants]
  Ascites | 14 | 14 | 28
  Bone | 168 | 162 | 330
  Breast | 61 | 63 | 124
  Chest Wall | 53 | 53 | 106
  Effusion | 57 | 55 | 112
  Lymph Node | 250 | 249 | 499
  Other | 20 | 18 | 38
  Peritoneum | 7 | 14 | 21
  Pleura | 29 | 35 | 64
  Skin/Soft Tissue | 60 | 62 | 122
  Visceral, Liver | 245 | 228 | 473
  Visceral, Lung | 180 | 174 | 354
  Visceral, Other | 34 | 28 | 62
Disease Sites at Baseline [Number; unit: participants]
  Liver ± Lung ± Skin/Soft Tissue ± Bone | 245 | 228 | 473
  Lung ± Skin/Soft Tissue ± Bone | 71 | 87 | 158
  Skin/Soft Tissue ± Bone | 49 | 52 | 101
  Bone | 0 | 3 | 3
  Other | 6 | 5 | 11
Karnofsky Performance Status [Number; unit: Units on a scale] — Karnofsky Performance Scale Index measures a patient's functional impairment: 100-80=Able to carry on normal activity and work, no special care; 70-50=Unable to work; able to live at home and care for most personal needs with assistance; 40-0=Unable to care for self; institutional or hospital care needed. Score reported in multiples of 10.
  Units on a scale
    100 | 108 | 105 | 213
    90 | 145 | 132 | 277
    80 | 86 | 102 | 188
    70 | 33 | 34 | 67
    <70 | 0 | 1 | 1
    Not reported | 3 | 3 | 6
Menopausal Status [Number; unit: participants]
  Premenopausal | 54 | 51 | 105
  Perimenopausal | 19 | 23 | 42
  Postmenopausal | 288 | 289 | 577
  Not reported | 14 | 14 | 28
Number of Disease Sites [Number; unit: participants]
  1 disease site | 39 | 34 | 73
  2 disease sites | 85 | 98 | 183
  3 disease sites | 110 | 121 | 231
  4 disease sites | 79 | 69 | 148
  ≥5 disease sites | 58 | 53 | 111
Presence of All Lesions [Number; unit: participants]
  Subjects with at least 1 lesion | 371 | 375 | 746
  Subjects with no lesions | 4 | 2 | 6
Visceral Disease in Liver and/or Lung [Number; unit: participants]
  Yes | 316 | 315 | 631
  No | 55 | 60 | 115
  Missing | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Per Independent Radiology Review Committee (IRRC)
Description: PFS defined as the time in months from randomization to date of progression. Patients who died without a reported prior progression were considered to have progressed on date of death; those who didn't progress or die were censored on date of last tumor assessment. Median PFS time with 95% CI estimated using the Kaplan Meier product limit method.
Time Frame: based on assessments every 6 weeks while on treatment until documented disease progression/unacceptable toxicity
Population: PFS was analyzed on all randomized patients on an intention to treat basis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ixabepilone + Capecitabine | Capecitabine
Number analyzed (Participants) | 375 | 377
Months | 5.85 [5.45 to 6.97] | 4.17 [3.81 to 4.50]
Statistical Analysis 1: Comparison: Ixabepilone + Capecitabine vs Capecitabine; Study required 615 events to achieve 90% power to detect a hazard ratio of 0.77 using a 2-sided α = 0.05 log-rank test. The analysis was a comparison between the 2 treatment arms using a 2-sided α=0.0483 log-rank test (adjusted for an interim analysis using the O'Brien Fleming spending function) to reject the null hypothesis of equality of progression free survival. The analysis was conducted when 639 events (310 in combination:329 in capecitabine) were observed from the 752 randomized patients; Test type: Superiority or Other; p = .0003, Log Rank — Test was stratified by 1) presence of visceral metastases in liver or lung, 2) minimum of either doxorubicin 420 mg/m2 or epirubicin 360 mg/m2, and relapse > 6 months in adjuvant setting, and 3) prior chemotherapy for metastatic disease. (yes/no); 95.17% confidence interval is adjusted for the interim analysis; Hazard Ratio (HR) = 0.75, 95.17% CI [0.64 to 0.88]

2. Secondary Outcome: Overall Response Rate (ORR) Per IRRC
Description: Participants with best response of "Complete" or "Partial" according to Response Evaluation Criteria in Solid Tumors (RECIST) a 4-item scale wherein complete response=disappearance of all target lesions and partial response=30% decrease in the sum of the longest diameter of target lesions
Time Frame: based on assessments every 6 weeks while on treatment until documented disease progression/unacceptable toxicity
Population: The analysis of ORR was conducted on all randomized patients on an intent to treat basis.
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Ixabepilone + Capecitabine | Capecitabine
Number analyzed (Participants) | 375 | 377
percent | 34.7 [29.9 to 39.7] | 14.3 [10.9 to 18.3]
Statistical Analysis 1: Comparison: Ixabepilone + Capecitabine vs Capecitabine; The study had 95 percent power to detect a significant difference in ORR if the true response rate was 32 percent in the combination arm and 20 percent in the capecitabine arm; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.15, 95% CI [2.20 to 4.50]

3. Secondary Outcome: Duration of Response Per IRRC
Description: Computed for all patients with a best response of "Partial" or "Complete" per RECIST (a 4-item scale as described in previous outcome measure), calculated from the time when these criteria were first met until the first date of documented progression or death.
Time Frame: based on assessments every 6 weeks while on treatment until documented disease progression/unacceptable toxicity
Population: Results for duration of response apply to only those subjects with a response (defined as complete or partial response).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone + Capecitabine | Capecitabine
Number analyzed (Participants) | 130 | 54
months | 6.4 [5.6 to 7.1] | 5.6 [4.2 to 7.5]

4. Secondary Outcome: Time to Response Per IRRC
Description: Time to response was summarized using descriptive statistics and was defined as the time from first dose of study treatment until measurement criteria were first met for Partial Response or Complete Response.
Time Frame: based on assessments every 6 weeks while on treatment until documented disease progression/unacceptable toxicity
Population: Results for time to response apply to only those subjects with a response (defined as complete or partial response)
Measure: Median (Full Range); unit: weeks
Arm/Group | Ixabepilone + Capecitabine | Capecitabine
Number analyzed (Participants) | 130 | 54
weeks | 11.7 [4.4 to 61.4] | 12.0 [4.3 to 41.9]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death. Participants who did not die at the time of the analysis were censored at the latest follow-up date. Median OS with 95% CI was estimated using the Kaplan Meier product limit method.
Time Frame: from date of randomization until death
Population: Overall survival was analyzed on all randomized patients on an intent to treat basis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ixabepilone + Capecitabine | Capecitabine
Number analyzed (Participants) | 375 | 377
Months | 12.9 [11.5 to 14.2] | 11.1 [10.0 to 12.5]
Statistical Analysis 1: Comparison: Ixabepilone + Capecitabine vs Capecitabine; Study required 631 deaths to achieve 80% power to detect a Hazard ratio of 0.8 using a 2-sided α = 0.05 log rank test. The analysis was a comparison between the 2 treatment arms using a 2-sided α=0.05 log-rank test to reject the null hypothesis of equality of survival. The analysis was conducted when 639 deaths (318 in combination:321 in capecitabine) were observed from the 752 randomized patients; Test type: Superiority or Other; p = 0.1936, Log Rank — Test was stratified by presence of visceral metastases in liver or lung (y/n), minimum of either doxorubicin 420 mg/m2 or epirubicin 360 mg/m2, and relapse > 6 months in adjuvant setting (y/n), and prior chemotherapy for metastatic disease (y/n); Test was conducted at the α=0.05 level and no adjustments were performed; Hazard Ratio (HR) = 0.90, 95.17% CI [0.77 to 1.05] — Confidence Interval adjusted for interim analysis

6. Secondary Outcome: Treatment-related Safety Summary
Description: Laboratory values, adverse events, and other symptoms were graded using the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTC) Version 3.0
Time Frame: safety was assessed on a continual basis every cycle while on-treatment and every 4 weeks post treatment until toxicities resolved or were deemed irreversible.
Population: All treated participants; all participants who received at least 1 dose of study therapy.Participants with baseline hepatic impairment (combination arm, n = 29; capecitabine arm, n = 35), defined as Grade ≥2 AST, ALT or Grade ≥1 total bilirubin, were contraindicated due to disproportionate number of toxic deaths.
Measure: Number; unit: Participants
Groups:
- Ixabepilone + Capecitabine: Ixabepilone in combination with capecitabine (combination group): Ixabepilone 40 mg/m2 administered as a 3-hour intravenous (IV) infusion on Day 1 of each cycle only, plus oral capecitabine 1000 mg/m2 twice a day (BID) (2000 mg/m2 daily dose) x 14 days, followed by 1 week of rest.
Arm/Group | Ixabepilone + Capecitabine | Capecitabine
Number analyzed (Participants) | 369 | 368
Participants
  Deaths on-study or within 30 days of last dose | 33 | 40
  Treatment-related Serious Adverse Events (SAEs) | 91 | 31
  Treatment-related Adverse Events (AEs) | 357 | 330
  Treatment-related AEs leading to Discontinuation | 137 | 25

7. Secondary Outcome: Symptom Assessment Score Changes From Baseline for Functional Assessment of Cancer Therapy-Breast Symptom Index (FBSI)
Description: Quality of life, as measured by the FBSI, an 8-item, participant-reported instrument to measure symptoms. Each item has 5 possible responses ranging from 0 (not at all) to 4 (very much). The scoring was conducted according to the Functional Assessment of Chronic Illness Therapy manual, Version 4; higher scores reflect fewer symptoms.
Time Frame: Baseline and prior to each 21-day cycle of treatment, and at first posttreatment follow-up assessment.
Population: Analysis was conducted on all randomized participants on an intent to treat basis.(Note: while table only reports data up to 24 wks, which represents most results, statistical analysis includes ALL assessments through study and follow-up; a few participants were assessed after more than 100 weeks.)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ixabepilone + Capecitabine | Capecitabine
Number analyzed (Participants) | 375 | 377
units on a scale
  Week 3 (n=282; n=273) | -0.4 [-0.97 to 0.20] | 0.3 [-0.28 to 0.84]
  Week 6 (n=227; n=214) | -0.2 [-0.90 to 0.48] | 1.1 [0.30 to 1.83]
  Week 9 (n=194; n=184) | -0.6 [-1.31 to 0.19] | 1.8 [0.97 to 2.58]
  Week 12 (n=173; n=158) | -1.3 [-2.19 to -0.42] | 1.4 [0.55 to 2.18]
  Week 15 (n=148; n=145) | -0.7 [-1.65 to 0.27] | 1.7 [0.73 to 2.72]
  Week 18 (n=122; n=121) | -1.0 [-2.18 to 0.13] | 1.7 [0.76 to 2.63]
  Week 21 (n=116; n=101) | -0.7 [-1.63 to 0.28] | 1.1 [0.01 to 2.21]
  Week 24 (n=95; n=82) | -0.8 [-1.89 to 0.38] | 2.3 [1.13 to 3.41]
Statistical Analysis 1: Comparison: Ixabepilone + Capecitabine vs Capecitabine; There was a statistically significant difference between groups in change from baseline FBSI score favoring capecitabine. A mean change from baseline of 2.5 was considered a clinically meaningful difference (minimally important difference or MID). On-treatment mean changes in the FBSI did not reach the MID in either group; Test type: Superiority or Other; p = .0002, Wei-Lachin

ADVERSE EVENTS:
Arm/Group | Capecitabine | Ixabepilone + Capecitabine
Serious Adverse Events (participants affected / at risk) | 127/368 | 151/369
Other Adverse Events (participants affected / at risk) | 350/368 | 360/369
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine (N=368) | Ixabepilone + Capecitabine (N=369)
HAEMOGLOBIN DECREASED (Investigations) | 1 | 1
GRIP STRENGTH DECREASED (Investigations) | 0 | 1
PLATELET COUNT DECREASED (Investigations) | 2 | 2
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 1
GRANULOCYTE COUNT DECREASED (Investigations) | 0 | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 1
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 0 | 1
CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 | 1
VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 3
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 2 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 0 | 1
THROMBOSIS (Vascular disorders) | 0 | 3
VASCULITIS (Vascular disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 2 | 3
LYMPHOEDEMA (Vascular disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 1
THROMBOPHLEBITIS (Vascular disorders) | 1 | 0
HYPOVOLAEMIC SHOCK (Vascular disorders) | 0 | 1
POOR VENOUS ACCESS (Vascular disorders) | 1 | 2
DEEP VEIN THROMBOSIS (Vascular disorders) | 4 | 0
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 0 | 1
DISORIENTATION (Psychiatric disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 2 | 2
HEPATIC FAILURE (Hepatobiliary disorders) | 4 | 1
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 1
HEPATOCELLULAR DAMAGE (Hepatobiliary disorders) | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 2
TYPE IV HYPERSENSITIVITY REACTION (Immune system disorders) | 0 | 1
APHASIA (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 1 | 1
HEADACHE (Nervous system disorders) | 1 | 1
LETHARGY (Nervous system disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 4
NEURALGIA (Nervous system disorders) | 0 | 1
CONVULSION (Nervous system disorders) | 2 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 1
PARAESTHESIA (Nervous system disorders) | 0 | 1
HYPOAESTHESIA (Nervous system disorders) | 0 | 1
MENTAL IMPAIRMENT (Nervous system disorders) | 0 | 1
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 | 1
COGNITIVE DISORDER (Nervous system disorders) | 1 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1
COORDINATION ABNORMAL (Nervous system disorders) | 1 | 1
INTERCOSTAL NEURALGIA (Nervous system disorders) | 1 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 2
PARESIS CRANIAL NERVE (Nervous system disorders) | 1 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 | 1
MARCHIAFAVA-BIGNAMI DISEASE (Nervous system disorders) | 1 | 0
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 | 3
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 5
ILEUS (Gastrointestinal disorders) | 1 | 3
NAUSEA (Gastrointestinal disorders) | 5 | 8
ASCITES (Gastrointestinal disorders) | 2 | 1
COLITIS (Gastrointestinal disorders) | 1 | 0
MELAENA (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 8 | 12
CHEILITIS (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 15 | 14
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1
ENTERITIS (Gastrointestinal disorders) | 2 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 1
STOMATITIS (Gastrointestinal disorders) | 1 | 3
CONSTIPATION (Gastrointestinal disorders) | 2 | 1
HAEMATEMESIS (Gastrointestinal disorders) | 1 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 0 | 1
PEPTIC ULCER (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 4
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0
EROSIVE OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL ULCER (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 2
SEPSIS (Infections and infestations) | 0 | 5
MYIASIS (Infections and infestations) | 1 | 0
CYSTITIS (Infections and infestations) | 0 | 1
INFECTION (Infections and infestations) | 2 | 1
PNEUMONIA (Infections and infestations) | 3 | 17
CELLULITIS (Infections and infestations) | 0 | 3
ERYSIPELAS (Infections and infestations) | 1 | 1
LARYNGITIS (Infections and infestations) | 0 | 1
PARONYCHIA (Infections and infestations) | 0 | 1
BACTERAEMIA (Infections and infestations) | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 1
HERPES ZOSTER (Infections and infestations) | 2 | 2
GASTROENTERITIS (Infections and infestations) | 1 | 2
LOBAR PNEUMONIA (Infections and infestations) | 0 | 1
PERITONEAL INFECTION (Infections and infestations) | 1 | 0
NEUTROPENIC INFECTION (Infections and infestations) | 0 | 1
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 0 | 1
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 0 | 1
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 2
GENITOURINARY TRACT INFECTION (Infections and infestations) | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0
ANOREXIA (Metabolism and nutrition disorders) | 2 | 2
DEHYDRATION (Metabolism and nutrition disorders) | 3 | 8
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 3
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 3
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 2
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 1
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 3 | 11
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 6
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 18
COAGULOPATHY (Blood and lymphatic system disorders) | 3 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 7
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 0 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 4 | 15
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 | 1
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 | 5
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 2
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
POST LUMBAR PUNCTURE SYNDROME (Injury, poisoning and procedural complications) | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 3
TRISMUS (Musculoskeletal and connective tissue disorders) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 3 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 2
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 | 14
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYDROTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 4 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 2
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 9 | 6
HYDROPNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 2
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 4
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PAIN (General disorders) | 0 | 2
DEATH (General disorders) | 1 | 2
CHILLS (General disorders) | 0 | 1
FATIGUE (General disorders) | 1 | 3
PYREXIA (General disorders) | 3 | 9
ASTHENIA (General disorders) | 2 | 3
CHEST PAIN (General disorders) | 1 | 1
SUDDEN DEATH (General disorders) | 0 | 1
GENERALISED OEDEMA (General disorders) | 1 | 0
MUCOSAL INFLAMMATION (General disorders) | 3 | 4
PERFORMANCE STATUS DECREASED (General disorders) | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 1
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTATIC PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
INFECTED NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MALIGNANT ASCITES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
METASTASES TO MENINGES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 36 | 19
PERICARDIAL EFFUSION MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 7
RENAL CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine (N=368) | Ixabepilone + Capecitabine (N=369)
LACRIMATION INCREASED (Eye disorders) | 21 | 21
WEIGHT DECREASED (Investigations) | 43 | 88
HAEMOGLOBIN DECREASED (Investigations) | 4 | 21
NEUTROPHIL COUNT DECREASED (Investigations) | 6 | 27
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 3 | 23
INSOMNIA (Psychiatric disorders) | 25 | 61
HEADACHE (Nervous system disorders) | 41 | 63
DIZZINESS (Nervous system disorders) | 36 | 48
DYSGEUSIA (Nervous system disorders) | 14 | 42
PARAESTHESIA (Nervous system disorders) | 22 | 71
HYPOAESTHESIA (Nervous system disorders) | 9 | 29
NEUROPATHY PERIPHERAL (Nervous system disorders) | 5 | 29
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 8 | 68
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 30 | 139
NAUSEA (Gastrointestinal disorders) | 164 | 209
VOMITING (Gastrointestinal disorders) | 106 | 158
DIARRHOEA (Gastrointestinal disorders) | 147 | 179
DYSPEPSIA (Gastrointestinal disorders) | 35 | 34
STOMATITIS (Gastrointestinal disorders) | 39 | 61
CONSTIPATION (Gastrointestinal disorders) | 57 | 120
ABDOMINAL PAIN (Gastrointestinal disorders) | 51 | 68
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 12 | 19
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 31 | 45
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 16 | 23
ANOREXIA (Metabolism and nutrition disorders) | 69 | 127
DECREASED APPETITE (Metabolism and nutrition disorders) | 8 | 21
ANAEMIA (Blood and lymphatic system disorders) | 10 | 19
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 22
NEUTROPENIA (Blood and lymphatic system disorders) | 9 | 51
RASH (Skin and subcutaneous tissue disorders) | 27 | 45
ALOPECIA (Skin and subcutaneous tissue disorders) | 16 | 121
DRY SKIN (Skin and subcutaneous tissue disorders) | 25 | 23
ERYTHEMA (Skin and subcutaneous tissue disorders) | 17 | 25
PRURITUS (Skin and subcutaneous tissue disorders) | 15 | 21
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 36 | 76
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 53 | 41
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 228 | 235
MYALGIA (Musculoskeletal and connective tissue disorders) | 24 | 130
BACK PAIN (Musculoskeletal and connective tissue disorders) | 53 | 46
BONE PAIN (Musculoskeletal and connective tissue disorders) | 19 | 26
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 25 | 87
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 30 | 70
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 16 | 41
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 20 | 20
COUGH (Respiratory, thoracic and mediastinal disorders) | 59 | 73
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 67 | 61
PAIN (General disorders) | 8 | 27
FATIGUE (General disorders) | 97 | 160
PYREXIA (General disorders) | 47 | 56
ASTHENIA (General disorders) | 57 | 101
CHEST PAIN (General disorders) | 19 | 22
OEDEMA PERIPHERAL (General disorders) | 46 | 51
MUCOSAL INFLAMMATION (General disorders) | 39 | 59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.